CLINICAL TRIAL: NCT02507518
Title: Role of 18FDG PET in the Evaluation of Early Response to Maintenance Treatment With Bevacizumab or Pemetrexed in Advanced Non-small-cell Lung Cancer
Brief Title: Role of PET Scan in the Evaluation of Early Response to Maintenance Treatment in Advanced Non-small-cell Lung Cancer
Acronym: CALMETTE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB12.01
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer, PET, progression free survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Two Pet scan Imaging will be done : 14 days before and 16 days after the beginning of maintenance therapy
  Interventions: Procedure: PET scan imaging

INTERVENTIONS:
Procedure: PET scan imaging — a PET scan will be done 2 weeks before the start of maintenance therapy and another 16 days after to predict the earlier response to treatment

SUMMARY:
Non small cell lung cancer is the first cause of cancer related death in France and is becoming an increasing health problem in developing countries.

Recently for patient with no progression disease after first line chemotherapy, new therapies were validated in maintenance (bevacizumab) or switch maintenance treatment (erlotinib, pemetrexed) with improved survival.

Until now, determination of efficiency of treatment is only based on morphological response (RECIST) and remains inappropriate to such cytostatic drugs for which there is no anatomical lesion modification.

Nuclear Medicine and especially 18-FDG Positron Emission Tomography (PET) offers a biologically relevant tool for assessment of tumour response therapies.

The assumption of the study is that FDG PET would allow to earlier detect a lack of response, thereafter, to modify an ineffective treatment. Indeed, nowadays the treatment is maintained up to evidence of progression disease.

However, despite the increasing use of FDG PET for predicting therapeutic response, there are no validated criteria for judging response of maintenance therapy in non-small cell lung cancer.

It seems necessary to determine standardized criteria response, earlier during the course of maintenance therapy in patient with non small cell lung cancer.

The final aim is to optimize survival by an adapted metabolic imaging guided therapy.

DETAILED DESCRIPTION:
The purpose of the study is to optimize survival by an adapted metabolic imaging therapy in patients with advances non-small cell lung cancer.

The primary objective of the study is to evaluate the role of SUV and metabolic volume measured by FDG PETScan in the early prediction of treatment response.

80 patients will be included in 2 years. They will be follow up for one year for monitoring the progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 years old
* Effective contraception method or negative pregnancy test at the inclusion
* OMS inferior or equal to 1
* Non-small cell lung cancer stage IIIb or IV
* Non progressive disease after at lest 4 cycles of platinum-based chemotherapy
* Eligible fo maintenance therapy with bevacizumab and/or pemetrexed
* Inform consent signed

Exclusion Criteria:

* Evolution of a second cancer in the 3 years before inclusion
* Pregnancy or breast-feeding
* poorly controlled diabetes
* curatorship or guardianship
* contraindication to iodinated contrast agents
* participation to another clinical research with an experimental drug
* impossible decubitus
* not possibility to follow-up the procedures of the study due to geographic, social or psychic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 16 weeks after the start of maintenance therapy
  time between the start of maintenance therapy and progression

SECONDARY OUTCOMES:
progression free survival | on year
  time between the start of maintenance therapy and progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Becker, MD, Principal Investigator — Centre Henri Becquerel
Locations (5):
- France (5):
  - CHU Rouen-Hôpital Bois-Guillaume, Bois-Guillaume
  - CH Dieppe, Dieppe
  - Centre hospitalier intercommunal Elbeuf Louviers, Elbeuf
  - Centre Henri Becquerel, Rouen
  - CHU Rouen, Rouen